CLINICAL TRIAL: NCT01018966
Title: Phase I Study of Ixabepilone (BMS-247550) in Patients With Solid Tumors
Brief Title: Study of Ixabepilone (BMS-247550) in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-029
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Solid Tumors
MeSH Terms: interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixabepilone (Experimental)
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Lyophilized and solvent, IV, 10-50 mg/m2, Q3W, At least 1 cycle, (21 days)
  Other Names: Ixempra; BMS-247550

SUMMARY:
The purpose of this study is to determine the DLT, MTD and recommended Phase II dose of ixabepilone in Japanese patients with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 20 years or older
* Histologically or cytologically confirmed diagnosis of adenocarcinoma Solid tumors

Exclusion Criteria:

* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≥2

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2004-04; Primary Completion 2005-03 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose (MTD), and a recommended Phase II dose of Ixabepilone when administered every three weeks by assessing status of treatment, dose intensity, and dose-limiting toxicities (DLT) | 3-week treatment cycles until unacceptable toxicity

SECONDARY OUTCOMES:
To evaluate safety by assessing adverse events. Toxicity will be evaluated according to the Common Toxicity Criteria Version 3.0 (CTC). Response will be evaluated according to the RECIST (Response Evaluation Criteria in Solid Tumors) criteria | 3-week treatment cycles
To evaluate the plasma pharmacokinetics of Ixabepilone according to the following parameters: Cmax, AUC(INF), Tmax, t1/2, MRT(INF), Vss, Cltot | Cycle 1 (first 3 weeks of study therapy)
To describe any preliminary evidence of anti-tumor activity (response), assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) | 3-week treatment cycles until unacceptable toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx